CLINICAL TRIAL: NCT03443986
Title: Effect of Resistance Training Associated With Whole-Body Vibration Over the Peripheral Circulation and the Functional Performance of the Elderly With Type 2 Diabetes: Randomized Controlled Clinical Trial
Brief Title: Effect of Resistance Training Associated With Whole-Body Vibration in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, Professor, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Resistance, Vibration and DM
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Blood Flow Velocity; Skin Temperature; Postural Balance; Combined Modality Therapy; Vibration; Resistance Training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: Three groups: resistance training associated with whole body vibration (G1), resistance training associated with vibration sham; (G2) and control group-guidelines about foot care (GC)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple: a researcher shall be exclusively responsible for the evaluations and reevaluations not having knowledge of what intervention
  group the patient will enter. The patient will be allocated among three groups. After the final evaluations, all data will be analyzed by another researcher directed solely to that purpose. Therefore, there will be a triple blinding (researcher, patient and statistician).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance training associated with vibration (Experimental): The workout will be held three times a week and will last a total of 12 weeks (3 months) for 45 minutes.
  Interventions: Other: Resistance training associated with vibration
- Resistance training associated with sham (Sham Comparator): The workout will be held three times a week and will last a total of 12 weeks (3 months) for 45 minutes, where there will be 5 minutes of heating, 19 minutes of exercise with load, 16 minutes of vibration "sham" and 5 minutes of slowdown. The vibration sham; will be held with the disconnected platform. A device will be connected producing a noise similar to the sound of the connected platform for a time equivalent to the treatment protocol, since it will not be possible to distinguishing noticeably stimulate vibrator. Participants that will undergo false vibration will not have contact with those who carry out the real treatment.
  Interventions: Other: Resistance training associated with vibration sham
- Control group (No Intervention): Will not be submitted to any physical intervention. It continues in your daily life with only monitoring via phone callings. Guidelines about foot care.

INTERVENTIONS:
Other: Resistance training associated with vibration — The workout will be held three times a week and will last a total of 12 weeks (3 months) for 45 minutes, where there will be 5 minutes of heating, 19 minutes of exercise with load, 16 minutes of vibration and 5 minutes of slowdown.
  Arms: Resistance training associated with vibration
Other: Resistance training associated with vibration sham — he workout will be held three times a week and will last a total of 12 weeks (3 months) for 45 minutes, where there will be 5 minutes of heating, 19 minutes of exercise with load, 16 minutes of vibration "sham" and 5 minutes of slowdown.
  Arms: Resistance training associated with sham

SUMMARY:
Introduction: Diabetes Mellitus (DM) is an important health condition of the population and its prevalence continues to grow due to population aging, economic development and urbanization. The exercise is an important factor of prevention and control, thereby decreasing the risk of metabolic diseases, cardiovascular diseases and improving the functionality of the patient with diabetes.

Objective: Evaluate the response of resistance training associated with whole-body vibration on peripheral circulation and functional performance of elderly with type 2 diabetes.

Methods: This is a clinical trial study, controlled, randomized and blinded, which will follow the guidelines established by the Consolidated Standards of Reporting Trials (CONSORT). Patients will be recruited in the light of the eligibility criteria and randomly divided into 3 groups: resistance training associated with whole body vibration (G1), resistance training associated with vibration sham (G2) and control group-guidelines about foot care (GC), establishing 36 treatment sessions, three times a week for the G1 and G2.

ELIGIBILITY:
Inclusion Criteria:

* Present overweight or obese class I, with BMI between 25.00 and 34.99 kg/m2 (WHO, 2009)
* Be functionally independent
* Having cognitive ability to respond and perform the exercisesevaluated by Mini-Mental State examination (MMSE), prepared by Folstein et al. (1975) and translation/modification proposed by Lawrence and van Heerden (2006), using as a bridge to cut to illiterate individuals = 19 points (BRAZIL, 2006)
* Inactive (0 to 5 points) or less active (6 to 11 points) according to the Questionnaire of Habitual Physical Activity (QAFH)
* Patients without severe foot deformities requiring therapeutic shoes
* Do not have orthopedic deficiencies
* No indications of deep vein thrombosis
* Do not use locomotion auxiliary equipment

Exclusion Criteria:

* Change in the drug program in during the research
* Performing other physical activity during the training
* Hypertensive Peaks during treatment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2020-04-08 (Estimated)

PRIMARY OUTCOMES:
Peripheral circulation | 12 weeks
  Vascular Doppler ultrasound (UVD)
Functional performance | 12 weeks
  Timed Up and Go Test (TUG)
Peripheral circulation | 12 weeks
  Infrared Thermography (TI)

SECONDARY OUTCOMES:
Static postural alignment | 12 weeks
  Optoeletrônico system SMART DX100
Plantar pressure distribution | 12 weeks
  Baropodometry

CONTACTS AND LOCATIONS:
Locations (1):
- François Talles Medeiros Rodrigues, Recife, Pernambuco, Brazil